CLINICAL TRIAL: NCT03230955
Title: Effectiveness of a Smoking Cessation Quit Line for Mental Health Patients: Pragmatic Clinical Trial
Brief Title: Effectiveness of a Smoking Cessation Quit Line for Mental Health Patients
Acronym: QUITMENTAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Català d'Oncologia (Other)
Collaborators: Hospital Universitari de Bellvitge (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Hospital Clinic of Barcelona (Other); Hospital Vall d'Hebron (Other); Hestia Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 061 QUIT_MENTAL PI15/00875
Record Dates: First submitted 2017-03-29; First posted 2017-07-27 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Mental Disorder; Smoking Cessation; Motivation
Keywords: Randomized clinical trial; Hotlines
MeSH Terms: conditions — Mental Disorders; Smoking Cessation | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into IG and CG with 2:1 allocation using mapping software, because it is expected a larger number of losses to follow-up in the CG. GI patients will be contacted by a nurse of the 061CatSalut Respon "quit line" who will have received specific training in intervening smokers with mental disorders. The call will take place within the first 48 h after discharge from the hospitals. The patients of the CG will be contacted by a team of the 061 CatSalut Respon in order to provide a brief counselling (first call) and evaluate their use of tobacco during the 1st, 6th and 12th month.
Who Masked: Participant
Masking Description: Participants and hospital clinicians will be blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychological and psycho-educational support (Experimental): The intervention group (IG) [that will receive telephone-based assistance to quit (including psychological and psycho-educational support and pharmacological treatment advice, if required) provided by trained nurses who will proactively call at one week, 15 day, a month, 3, 6 and 12 months after discharge, plus the calls made by the patients during the process]
  Interventions: Behavioral: Psychological and psycho-educational support by phone
- Control Group (Active Comparator): The control group (CG) [that will receive only a brief counselling session after discharge]
  Interventions: Other: Brief counselling session

INTERVENTIONS:
Behavioral: Psychological and psycho-educational support by phone — The intervention is based on cognitive-behavioural therapy (CBT). The intervention, in order to achieve behavioural changes, will include components based in Bandura's social learning theory and social cognitive theory (Bandura, 1986) and the transtheorical model of change (Prochaska, 1992). It has been shown that expectations and self-efficacy are behavioural predictors and that they are an effective framework for the assistance to quit smoking. This theory allows evaluating patient motivation phase and adapting the interventions according to each phase (Fiore, 2011)
  Other Names: Telephone-based motivational intervention
  Arms: Psychological and psycho-educational support
Other: Brief counselling session — Brief counselling session
  Other Names: Brief advice
  Arms: Control Group

SUMMARY:
Pragmatic randomized clinical trial, single-blind, with allocation 2:1 [Intervention Group (IG) and control group (CG)] in 5 acute hospitals. The IG will receive telephone assistance to quit smoking (including psychological and psycho-educational support and pharmacological treatment advice, if required) proactively for 12 months, and the CG only brief counselling after discharge.

To assess the effectiveness of a multicomponent and motivational intensive telephone-based intervention to stop smoking ("quit line") addressed to smokers with mental disorders discharged from hospitals.

DETAILED DESCRIPTION:
Background: People suffering from mental illness are more likely to smoke. In Spain, up to 75% of patients hospitalized for mental disorders smoke, tripling the general population consumption. Life expectancy for people with severe mental illnesses is decreased by up to 25 years in comparison to the general population, mainly due to diseases caused or worsened by smoking. Hospitalized patients without monitoring after discharge quickly restore their tobacco use to previous levels. This evidence suggests the need of an appropriate follow-up intervention to prevent relapse after discharge and achieve higher rates of withdrawal in this population.

Objectives: To assess the effectiveness of a multicomponent and motivational intensive telephone-based intervention to stop smoking ("quit line") addressed to smokers with mental disorders discharged from hospitals.

Methods: Pragmatic randomized clinical trial, single-blind, with allocation 2:1 [Intervention Group (IG) and control group (CG)] in 5 acute hospitals. The IG will receive telephone assistance to quit smoking (including psychological and psycho-educational support and pharmacological treatment advice, if required) proactively for 12 months, and the CG only brief counselling after discharge. The sample size, calculated with an expected difference of 15 points on withdrawal between groups, α=0.05 and β=0.10 and 20% loss, will be of 334 (IG) and 176 (CG), which will be doubled to allow stratified analyses. Variables: a) dependent variables: self-reported smoking abstinence and verified by expired carbon monoxide levels, quit attempts, time of abstinence, motivation and self-efficacy to quit, and b) independent variables: age, sex and main disorder. Data analysis: multivariate logistic regression (odds ratio and confidence interval, CI 95%) of abstinence and other variables adjusted for potential confounding variables. Number of smokers needed to treat (NNT, and its 95% CI) to achieve one abstinent will be calculated.

Hypothesis: Abstinence rate (≥ 15%) of enrolled patients between groups. If the intervention is effective, the pragmatic nature of the study will permit to transfer it to the routine clinical practice with a reasonable investment.

ELIGIBILITY:
Inclusion Criteria:

1. smokers;
2. adults of both sexes ≥ 18 years to ≤76 years of age;
3. that have stayed in an Acute or Detoxification mental health unit for more than 24 hours;
4. with a telephone, fixed or mobile;
5. residents in the metropolitan area of Barcelona;
6. that provide their informed consent.

Exclusion Criteria:

1. patient discharged from the psychiatric emergency room;
2. with dementia or brain damage;
3. that do not speak Spanish or Catalan;
4. pregnant women;
5. with hearing and/or speech deficit;
6. with insufficient reading comprehension skills in Spanish or Catalan;
7. that are trying to quit in smoking in another centre, or using another intervention in that moment;
8. that have voluntarily requested discharge;
9. that plan to shift their domicile outside of Barcelona county.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change from tobacco consumption abstinence at 12 months | through study completion, an average of 1 year
  Tobacco consumption abstinence (yes/no), self-reported the day of recruitment and 12 months after discharge (7 days abstinence prior to the evaluation point)

SECONDARY OUTCOMES:
Change in the level of self-efficacy to quit smoking | through study completion, an average of 1 year
  Change of self reported self-efficacy (using a Likert scale from 0 to 10)
Change of motivation to quit smoking (stage of change) | through study completion, an average of 1 year
  The Stages of Change Model helps to know the patient's motivation to quit, or stage of change, in order to allow clinicians to tailor interventions according to each stage (Prochaska, 1992).
Attempts to quit smoking | through study completion, an average of 1 year
  Number of serious quit attempts after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Martínez, RN,BA, PhD, Principal Investigator — Institut Català d'Oncologia
Locations (1):
- Hospital Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared with other researchers

REFERENCES:
- [Background] Ballbe M, Martinez C, Salto E, Cabezas C, Riccobene A, Valverde A, Gual A, Fernandez E. Maintenance of tobacco cessation programmes in public hospitals in Catalonia, Spain. Addict Behav. 2015 Mar;42:136-9. doi: 10.1016/j.addbeh.2014.11.028. Epub 2014 Nov 26. PMID 25462661
- [Background] Ballbe M, Nieva G, Mondon S, Pinet C, Bruguera E, Salto E, Fernandez E, Gual A; Smoking and Mental Health Group. Smoke-free policies in psychiatric services: identification of unmet needs. Tob Control. 2012 Nov;21(6):549-54. doi: 10.1136/tobaccocontrol-2011-050029. Epub 2011 Sep 20. PMID 21933940
- [Background] Ballbe M, Sureda X, Martinez-Sanchez JM, Salto E, Gual A, Fernandez E. Second-hand smoke in mental healthcare settings: time to implement total smoke-free bans? Int J Epidemiol. 2013 Jun;42(3):886-93. doi: 10.1093/ije/dyt014. Epub 2013 Mar 29. PMID 23543600
- [Background] Ballbe M, Sureda X, Martinez-Sanchez JM, Fu M, Salto E, Gual A, Fernandez E. Secondhand smoke in psychiatric units: patient and staff misperceptions. Tob Control. 2015 Oct;24(e3):e212-20. doi: 10.1136/tobaccocontrol-2014-051585. Epub 2014 Sep 19. PMID 25239470
- [Background] Banham L, Gilbody S. Smoking cessation in severe mental illness: what works? Addiction. 2010 Jul;105(7):1176-89. doi: 10.1111/j.1360-0443.2010.02946.x. Epub 2010 May 11. PMID 20491721
- [Background] Chabrol H, Niezborala M, Chastan E, de Leon J. Comparison of the Heavy Smoking Index and of the Fagerstrom Test for Nicotine Dependence in a sample of 749 cigarette smokers. Addict Behav. 2005 Aug;30(7):1474-7. doi: 10.1016/j.addbeh.2005.02.001. PMID 16022945
- [Background] Fiore MC, Baker TB. Clinical practice. Treating smokers in the health care setting. N Engl J Med. 2011 Sep 29;365(13):1222-31. doi: 10.1056/NEJMcp1101512. PMID 21991895
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Hughes JR, Keely JP, Niaura RS, Ossip-Klein DJ, Richmond RL, Swan GE. Measures of abstinence in clinical trials: issues and recommendations. Nicotine Tob Res. 2003 Feb;5(1):13-25. PMID 12745503
- [Background] Martinez C, Fu M, Martinez-Sanchez JM, Ballbe M, Puig M, Garcia M, Carabasa E, Salto E, Fernandez E. Tobacco control policies in hospitals before and after the implementation of a national smoking ban in Catalonia, Spain. BMC Public Health. 2009 May 28;9:160. doi: 10.1186/1471-2458-9-160. PMID 19473549
- [Background] Martinez C, Guydish J, Le T, Tajima B, Passalacqua E. Predictors of quit attempts among smokers enrolled in substance abuse treatment. Addict Behav. 2015 Jan;40:1-6. doi: 10.1016/j.addbeh.2014.08.005. Epub 2014 Aug 27. PMID 25218064
- [Background] Morris CD, Tedeschi GJ, Waxmonsky JA, May M, Giese AA. Tobacco quitlines and persons with mental illnesses: perspective, practice, and direction. J Am Psychiatr Nurses Assoc. 2009 Feb;15(1):32-40. doi: 10.1177/1078390308330050. PMID 21665792
- [Background] Morris CD, Waxmonsky JA, May MG, Tinkelman DG, Dickinson M, Giese AA. Smoking reduction for persons with mental illnesses: 6-month results from community-based interventions. Community Ment Health J. 2011 Dec;47(6):694-702. doi: 10.1007/s10597-011-9411-z. Epub 2011 May 10. PMID 21556784
- [Background] Prochaska JJ, Hall SE, Delucchi K, Hall SM. Efficacy of initiating tobacco dependence treatment in inpatient psychiatry: a randomized controlled trial. Am J Public Health. 2014 Aug;104(8):1557-65. doi: 10.2105/AJPH.2013.301403. Epub 2013 Aug 15. PMID 23948001
- [Background] Twyman L, Bonevski B, Paul C, Bryant J. Perceived barriers to smoking cessation in selected vulnerable groups: a systematic review of the qualitative and quantitative literature. BMJ Open. 2014 Dec 22;4(12):e006414. doi: 10.1136/bmjopen-2014-006414. PMID 25534212
- [Derived] Ballbe M, Martinez C, Feliu A, Torres N, Nieva G, Pinet C, Raich A, Mondon S, Barrio P, Hernandez-Ribas R, Vicens J, Costa S, Vilaplana J, Alaustre L, Vilalta E, Blanch R, Subira S, Bruguera E, Suelves JM, Guydish J, Fernandez E. Effectiveness of a telephone-based intervention for smoking cessation in patients with severe mental disorders: study protocol for a randomized controlled trial. Trials. 2019 Jan 11;20(1):38. doi: 10.1186/s13063-018-3106-5. PMID 30635072